CLINICAL TRIAL: NCT01478243
Title: Study of Psycho-Social Impact of Keloid
Status: Terminated | Type: Observational
Why Stopped: Lack of institutional support and IRB related issues.
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 11-07
Record Dates: First submitted 2011-11-20; First posted 2011-11-23 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Keloid
Keywords: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite their benign nature, keloids may constitute a severe aesthetic, and in some cases, functional problem which translates to various repercussions on person's quality of life, including much stress and insecurities.

Keloids are mostly observed between the ages of 10 and 30. Although keloid is a common condition and the investigators can make assumptions about those living with keloids, the investigators do not know the actual impact of the illness on the overall performance of patients' and how this disease, day to day, is impacting their lives. The investigators are conducting this study, aimed to investigate the psychosocial impact of keloid on daily life. Information is collected anonymously. You must be 18 years of age or older to take this survey. Parents can respond on behalf of their children who are not 18 years of age yet. The online survey will take 20-30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of Keloid
2. Informed consent
3. Age above 18 to answer the survey questions
4. Parents shall respond on behalf of their minor children

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with clinical diagnosis of Keloid are invited to particiapate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Principal Investigator — Keloid Research Foundation
Locations (1):
- Michael H. Tirgan MD, New York, New York, United States